CLINICAL TRIAL: NCT06263855
Title: Effect of Large Language Model in Assisting Discharge Summary Notes Writing for Hospitalized Patients: A Pilot Pragmatic Randomized Controlled Trial
Brief Title: Effect of Large Language Model in Assisting Discharge Summary Notes Writing for Hospitalized Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are no longer going to evaluate the intervention.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiaoxi Yao, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-000352
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Large Language Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clinicians who care for patients randomized to intervention will have access to CURE to assist with discharge summary writing.
  Interventions: Other: CURE
- Control (No Intervention): Clinicians who care for patients randomized to control will continue with standard practice for discharge summary writing.

INTERVENTIONS:
Other: CURE — A large language model (LLM) to help clinicians prepare discharge summaries for hospitalized patients.
  Arms: Intervention

SUMMARY:
This pilot study aims to assess the feasibility of carrying out a full-scale pragmatic, cluster-randomized controlled trial which will investigate whether discharge summary writing assisted by a large language model (LLM), called CURE (Checker for Unvalidated Response Errors), improves care delivery without adversely impacting patient outcomes.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Adult patients admitted to one of three participating cardiology services at Mayo Clinic in Rochester, MN

Exclusion Criteria:

* Minor patients (<18)
* Patients admitted to a hospital service where CURE is not implemented

CLINICIANS

Inclusion Criteria:

* Clinicians who provide care to randomized patients included in this pilot

Exclusion Criteria:

* Clinicians who do not provide care to randomized patients included in this pilot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patient accrual | Three months
  The first feasibility outcome will be the rate of patient accrual. An accrual of one patient per day will be considered acceptable, i.e., 91 patients discharged from a 91-day period who are appropriately randomized and can be included in the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Yao, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No